CLINICAL TRIAL: NCT06082180
Title: A Prospective, Open-label, Multicenter, Randomized Controlled Phase III Study of Prophylactic Central Neck Dissection in Low-risk Papillary Thyroid Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, liu jie, clinical professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAM
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Cancer; Recurrence
Keywords: Thyroid cancer; prophylactic central neck dissection; recurrence; thyroglobulin
MeSH Terms: conditions — Thyroid Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: test group: prophylactic central neck dissction; control group: no central neck dissection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): prophylactic central neck dissection
  Interventions: Procedure: prophylactic central neck dissection
- control group (No Intervention): no central neck dissection

INTERVENTIONS:
Procedure: prophylactic central neck dissection — prophylactic central neck dissection was performed for the ipsilateral lesion
  Arms: test group

SUMMARY:
papillary thyroid carcinoma (PTC) is the most common thyroid cancer and has a good prognosis. Surgery is the primary treatment for PTC, and occult lymph node metastasis is not uncommon (20%-80%).The lymph node metastasis of PTC is mostly along the lymphatic drainage path station by station, and most of the first metastasis is to the central lymph node. According to the 2015 American Thyroid Association recommendation, prophylactic central lymph node dissection is recommended for patients with primary T3-4 or cN1b without central lymph node involvement. However, PTC with primary site T1-2, no external invasion and cN0 could not be dissected by central lymph node.Previous studies have suggested that prophylactic dissection should be performed to improve disease-specific survival, reduce local recurrence, improve recurrence risk and treatment response assessment, and help RAI decision making. Although routine prophylactic central lymph node dissection may detect occult lymph node metastasis, the need for further dissection of the recurrent laryngeal nerve and the parathyroid gland may lead to an increased incidence of complications, while its effect on reducing the risk of recurrence and improving prognosis is unclear, and the impact on long-term outcomes may be small.Previous retrospective studies in our institution have shown that routine central neck dissection does not significantly reduce the risk of recurrence. This study was designed to evaluate the benefits and risks of prophylactic central lymph node dissection in cT1b-T2N0 patients with papillary thyroid carcinoma. In order to ameliorate the effects of relapse and long time of death of PTC, thyroglobulin and its antibodies were also evaluated for short-term treatment response after surgery.

ELIGIBILITY:
Inclusion Criteria:

- (1)Patients age 18-70 years old, ECOG score 0-2; (2)Thyroid nodule measuring 11-40 mm on ultrasound (cT1bT2) and with fine-needle aspiration biopsy (FNAB) cytology in favor of "papillary thyroid carcinoma" or with intraoperative frozen section analysis "papillary thyroid carcinoma" .

(3)cN0: absence of lymph nodes suspicious for malignancy on preoperative ultrasound performed by the center's designated radiologist according to a standardized report, no gross extrathyroidal extension was found before or during the surgery; (4)No serious medical disease and dysfunction of major organs, such as blood routine, liver, kidney, heart, and lung function; no previous history of other head and neck malignancies, no history of neck radiation, no history of deep neck surgery (skin mass resection except clinical); (5)Patients should understand, sign and date the written informed consent form prior to any protocol specific procedures. Patients should be able and willing to comply with study visits.

Exclusion Criteria:

-(1)History of malignancy in other sites (previous or concurrent), excluding curable non-melanoma skin cancer and cervical carcinoma in situ; (2)Tumors > 40 mm (cT3) or ≤ 10 mm; tumors with extrathyroidal extension suspected or obvious on the pre-operative work-up or intra-operatively; (3)Metastatic neck lymph nodes or suspicious neck nodes on preoperative ultrasound (cN1); for suspicious nodes, FNAB cytology and thyroglobulin assay on the needle washout fluid will be performed.Metastatic neck lymph nodes found during the thyroidectomy and confirmed with intra-operative frozen section analysis.

(4)No papillary thyroid carcinoma on FNAB cytology and/or high-risk subtype PTC; (5)Pregnant or breast feeding women (6)Participation in another therapeutic clinical trial within four months from study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1199 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
excellent response | 1 year
  To assess the effect of prophylactic central neck dissection for excellent response of cN0 low-risk papillary thyroid cancer

SECONDARY OUTCOMES:
recurrence-free survival | 1 year; 2 year
  to assess the influence of prophylactic central neck dissection on imporvement of RFS of cN0 low-risk papillary thyroid cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No